CLINICAL TRIAL: NCT00187304
Title: Anticoagulation Treatment Influence on Post-operative Patients -Action SJM EPIC Trial
Brief Title: ACTION - Anticoagulation Treatment Influence on Post-operative Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study replaced by an observational study
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS04012TV
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Valve Disease
MeSH Terms: conditions — Heart Valve Diseases | interventions — Transcatheter Aortic Valve Replacement

INTERVENTIONS:
Device: Aortic valve replacement

SUMMARY:
The primary objective of this study is to compare two different regimens of therapy, AVK and ASA (aspirin), in the early postoperative period after aortic valve replacement with SJM Epic™ or SJM Epic™ Supra Porcine Bioprosthetic Heart Valve by establishing the adverse event free survival rate at 3 month post intervention follow-up of the 2 groups(with special focus on thromboembolic events and bleedings).

ELIGIBILITY:
Inclusion Criteria:

1. Patient requires, for the first time, isolated aortic valve replacement (pacemaker insertion is allowed)
2. Patient (or legal guardian) has signed a study specific informed consent form agreeing to the data collection and follow-up requirements.
3. Patient is of legal age in the host country
4. The patient is in sinus rhythm before implantation

Exclusion Criteria:

1. Patient already has a prosthetic valve, other than the valve being replaced at this time.
2. Patient requires double valve implantation
3. Patient requires concomitant CABG
4. Patients requires intra aortic balloon pump at intervention
5. Patient has a medical condition which contraindicates implantation of the SJM Epic and/or SJM Epic Supra Porcine Bioprosthetic Heart Valve (e.g. patient on dialysis)
6. Patient requires ASA or AVK therapy, i.e. not suitable for randomization
7. Patient is pregnant or nursing.
8. Patient is affected by active endocarditis.
9. Patient is affected by aortic dissection.
10. Patient has history of cerebral ischemia
11. Patient is affected by coagulopathy, history of GI bleeding or increased bleeding risk
12. Patient is affected by peripheral vascular disease requiring treatment
13. Patient has previous chronic anticoagulation therapy
14. Patient is allergic to ASA and/or AVK

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Phillippe Verhoye, MD, Principal Investigator — CHU Pontchaillou Rennes France